CLINICAL TRIAL: NCT05814952
Title: An Open Label Dose Escalation Clinical Trial to Evaluate the Safety and the Efficacy of LX103 in Patients With X-Linked Retinoschisis (XLRS)
Brief Title: Safety and Efficacy Study of LX103 Treatment of X-Linked Retinoschisis (XLRS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Innostellar Biotherapeutics (Unknown)
Responsible Party: Principal Investigator, Xiaodong Sun, PhD, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHGH-LX103
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: X-linked Retinoschisis
MeSH Terms: conditions — Retinoschisis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LX103 Injection (Experimental): Potential doses:
  5E10 vg, 0.1 mL/eye/dose (low dose)
  1E11 vg, 0.05 mL/eye/dose (high dose)
  Interventions: Genetic: LX103 Injection

INTERVENTIONS:
Genetic: LX103 Injection — Qualified subjects will receive a single unilateral intravitreal injection of LX103 at Day 0 in the trial.

SUMMARY:
The goal of this study is to evaluate the safety and efficacy of LX103 treatment of X-linked retinoschisis. This study will enroll subjects aged ≥ 6 years old to receive a single unilateral intravitreal (IVT) injection of LX103 to evaluate its safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign the informed consent, and willing to attend follow-up visits.
2. Male individual at least 6 years of age with a diagnosis of XLRS and documented mutations in the RS1 gene.
3. The study eye must have a best-corrected E-ETDRS visual acuity letter score of less than or equal to 63.

Exclusion Criteria:

1. Any eye with disease that would interfere with the fundus examinations.
2. The study eye is receiving topical carbonic anhydrase inhibitor, or has received topical carbonic anhydrase inhibitors in the past three months.
3. The study eye has undergone intraocular surgery within six months prior to enrollment.
4. Participant has uncontrolled hypertension or diabetes.

Min Age: 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | 24 weeks
  Incidence of adverse events (AEs) within 24 weeks of LX103 intravitreal injection at different doses
Incidence of serious adverse events (SAEs) | 24 weeks
  Incidence of serious adverse events (SAEs) within 24 weeks of LX103 intravitreal injection at different doses

SECONDARY OUTCOMES:
Mean change from baseline in BCVA (LogMAR) in the study eye | 24 weeks, 52 weeks
  ETDRS visual acuity charts will be used to assess BCVA
Mean change from baseline in central subfield thickness (CST) in the study eye | 24 weeks, 52 weeks
  Mean change of CST measured using Optical Coherence Tomography (OCT)
Change from baseline in Electroretinogram (ERG) parameters in the study eye | 24 weeks, 52 weeks
  Change in dark-adapted 3.0 B-wave amplitude (μV)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No